CLINICAL TRIAL: NCT02008071
Title: Effects of a Minimal-Contact Lifestyle Intervention on Physical Activity, Diet, and Body Weight
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTK-123
Record Dates: First submitted 2013-11-13; First posted 2013-12-11 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2013-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily step goal financial incentive (Experimental)
  Interventions: Behavioral: Daily step goal financial incentive
- Control, Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Daily step goal financial incentive — Participants' daily activity was incentivized. Reaching a predetermined/individualized step goal each day resulted in 1.00 per day.
  Arms: Daily step goal financial incentive
Behavioral: Standard of Care — Standard payment of 70.00 at the beginning of the study. Participants' daily activity was not incentivized.
  Arms: Control, Standard of Care

SUMMARY:
The purpose of this study is to conduct a pilot randomized controlled trial, to determine whether providing financial incentives for meeting daily step goals (a) increases the daily step counts of participants, (b) increases compliance with the overall program (including diet recommendations), and (c) increases weight loss.

ELIGIBILITY:
Inclusion Criteria:

* required to be able to read.
* required to have access to a computer.
* required to have a body mass index between 27 and 45 kg.m-2.
* required to take fewer than 7,000 steps per day at baseline (as determined by a pedometer, averaged across 4-7 days).

Exclusion Criteria:

* Individuals who report having an injury or physical limitation that renders them unable to walk ¼ mile without difficulty.
* Uncontrolled cardiovascular or metabolic condition determined by health history questionnaire.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Daily Step Count | Change from week 1 to week 12
  Change in steps/day from week 1 to week 12.

SECONDARY OUTCOMES:
Program Compliance | Change from week 1 to week 12
  Compliance with the physical activity prescription, means meeting or exceeding the step goal for that day. Participants' compliance was assessed by totaling the number of days they met their step goal and dividing it by the total number of days of the intervention. Thus, providing investigators the percentage of days that each participant complied with their physical activity prescription.

OTHER OUTCOMES:
Weight Loss | Change from week 1 to week 12. There will also be measures taken 3 months following week 12
  Change in weight, waist circumference, and hip circumference from week 1 to week 12. There will also be measures taken 3 months following week 12. This will be defined as the follow-up data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States